CLINICAL TRIAL: NCT05440292
Title: Effects of Individualized Accurate Positioning TMS Based on Task fMRI Activation on Upper Extremity Function After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Xiao Lu
Record Dates: First submitted 2022-06-19; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging; Upper Extremity Dysfunction; Brain Plasticity
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hotspot-rTMS Group (Experimental): rTMS stimulate on the hotspot of unaffected hemisphere
  Interventions: Device: Transcranial magnetic stimulation
- fMRI-rTMS Group (Experimental): rTMS stimulate on the motor task activation poin (targeted by fMRI) of unaffected hemisphere
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — For each stimulation day, low-frequency (1 Hz) ,1800 pulses(intensity of 100% resting motor threshold(RMT), duration 30 min) rTMS stimulation were delivered on the hotspot of unaffected hemisphere(Hotspot-rTMS Group) and the motor task activation poin of unaffected hemisphere(fMRI-rTMS Group). rTMS which guided by individualized navigation delivery 5 days a week for 4 weeks.

SUMMARY:
Stroke is a global health problem and a leading cause of disability. Limitation of upper limb function occurs in 55 -75% of patients after stroke. In recent years, non-invasive brain stimulation techniques, such as repetitive transcranial magnetic stimulation (rTMS), have been shown that can promote functional recovery in stroke patients, and multiple studies have reported that low-frequency rTMS stimulation on the motor areas of the unaffected hemispheres of stroke patients can significantly improve motor function of the affected upper limb. The standard procedure for TMS to determine the primary motor area is to measure hotspot, which is used as a common target for movement disorders such as hemiplegia after stroke. In the 1990s, the hands-on task activation point determined by functional magnetic resonance imaging(fMRI) and positron emission computed tomography(PET) studies was located at "Hand Knob" in the primary motor area. The study found that although the hands-on task activation point was closer to hotspot, it was significantly different from hotspot. The hands-on task activation point had stronger functional connection with the whole brain, especially the motor cognition-related brain area. Therefore, this study aims to compare the efficacy of rTMS stimulation on individual rTMS targets(task fMRI activation point) with traditional hotspot in patients with post-stroke hemiplegia. The regulation effect of rTMS was evaluated by using local brain function indicators and functional connections, and the longitudinal change pattern of brain function before and after treatment was observed to explore the therapeutic targets of rTMS for motor dysfunction after stroke and the mechanism of brain functional plasticity.

ELIGIBILITY:
Inclusion Criteria:

1. patients with ischemic stroke;
2. Primary onset, non-lateral motor area stroke lesion, duration of disease 15 days to 1 year;
3. Hemiplegia with unilateral hemispheric injury;
4. Brunnstrom grading (Brunnstrom, 1966)≤ STAGE IV;
5. Unconscious disorder;
6. Can cooperate to complete scale assessment, MRI scan and TMS treatment;
7. Can complete manual tasks and obtain activation points in the lateral motor area of the healthy hemisphere;
8. The head movement amplitude of all fMRI images was translational < 2mm and rotational < 2°;
9. Consent to rTMS treatment on the basis of conventional treatment and pass TMS safety screening;

Exclusion Criteria:

1. Use of muscle relaxation drugs recently;
2. A history of epilepsy;
3. History of other neuropsychiatric diseases;
4. Other motor system diseases;
5. History of head trauma and serious heart disease;
6. Contraindications to MRI scanning (implantable pacemaker, cardiac catheter or electronic pump; Intracerebral metal aneurysm clip, metal nail or vascular suture device; Intracerebral nerve stimulator or brain/subdural electrode, etc.)
7. Skull defect was closed with metal plate at TMS stimulation site;
8. Patients with skull defect;
9. Other severe systemic diseases or clinical critical conditions (respiratory or hemodynamic instability);
10. Refuse to participate in the trial.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity | At the end of 4 weeks of rTMS
  Only scoring for the upper limb motor function, including 33 items, scores range from 0 to 66 points. The higher scores, the better upper limb function.
Fugl-Meyer Assessment-Upper Extremity Scale | 2 months after the end of rTMS
  Only scoring for the upper limb motor function, including 33 items, scores range from 0 to 66 points. The higher scores, the better upper limb function.

SECONDARY OUTCOMES:
Action Research Arm Test | At the end of 4 weeks of rTMS; 2 months after the end of rTMS
  Including 19 items, scores range from 0 to 57 points. The higher scores, the better upper limb function.
National Institute of Health Stroke Scale | At the end of 4 weeks of rTMS; 2 months after the end of rTMS
  Use for evaluating the severity of neurological impairment in stroke,including 11 items, scores range from 0 to 42 points. The higher scores, the more severe the neurological impairment.
Barthel Index | At the end of 4 weeks of rTMS; 2 months after the end of rTMS
  Use for evaluating the ability in activity of daily living, including 10 items,scores range from 0 to 100 points. The higher scores, the better ability in activity of daily living.
Regional homogeneity (ReHo), Amplitude of low-frequency fluctuation (ALFF), Functional connectivity (FC) | At the end of 4 weeks of rTMS; 2 months after the end of rTMS
  Resting state functional magnetic resonance scan.The increase of ReHo represents the enhancement of the consistency of spontaneous neural activity in local brain regions. The increase of ALFF represents the enhancement of spontaneous neural activity. The increase of FC represents the enhancement functional connectivity between different regions of brain.
Latency of motor evoked potential, Amplitude of motor evoked potential | At the end of 4 weeks of rTMS; 2 months after the end of rTMS
  The higher values of latency of motor evoked potential indicate the lower activity of motor cortex in brain. The higher values of amplitude of motor evoked potential indicate the higher activity of motor cortex in brain.
Surface electromyogram measurement | At the end of 4 weeks of rTMS; 2 months after the end of rTMS
  The affected side of the biceps brachii, triceps brachii, flexor carpi and extensor carpi dorsi. The higher values of root-mean-square and integrated electromyogram indicate the stronger muscle's ability to contract.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No